CLINICAL TRIAL: NCT03304977
Title: Current Situation of the Patient's Knowledge on Their Anticoagulating and Anti Platelet Treatment in GHPSJ (St Joseph's Hospital)
Brief Title: Patient's Knowledge on Their Anticoagulating and Anti Platelet Treatment St Joseph's Hospital)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CACHACA
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-09

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire via smartphone — questionnaire via smartphone

SUMMARY:
Oral antigoagulant are used more than 60 years in thrombotic diseases. Even they are indispensable, the haemorragic risk is high.That's why it's the main reason of hospitalization for iatrogeny.The complication's reasons are mainly linked to errors of drug intake, drugs interaction and the lack of understanding the treatment.Moreover, the antiplatelet agglutening treatment is frequently added to anticoagulant treatment.This increases the haemorragic risk.Different means were used to minimize the risk , like INR follow up.

The purpose of the study is to evaluate smartphone use to follow the patients'treatment.

DETAILED DESCRIPTION:
Two questionnaire via smartphone with 15 days gap.

ELIGIBILITY:
Inclusion Criteria:

* patient under ant-thrombotic treatment
* hospitalized in vascular medecine service

Exclusion Criteria:

* refusing the participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
smartphone use level | 15 days
  evaluation of the interest of patient to use their smartphone in the purpose to follow their anticoagulant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PRIOLLET, MD, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France